CLINICAL TRIAL: NCT01505595
Title: Proprioceptive Training and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr. Simon Brumagne, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012_SBrumagne_PT-LBP; 1.5.104.03, G.0674.09 (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Proprioceptive Training; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proprioceptive training (Experimental)
  Interventions: Other: Proprioceptive training
- Sham proprioceptive training (Sham Comparator)
  Interventions: Other: Sham proprioceptive training

INTERVENTIONS:
Other: Proprioceptive training — 12 weeks
  Arms: Proprioceptive training
Other: Sham proprioceptive training — Three times daily inspiratory muscle training (2x30 breaths) at an intensity of 10% Pi,max
  Arms: Sham proprioceptive training

SUMMARY:
Proprioceptive weighting changes may explain differences in postural control performance. Deficits in proprioception are found in a subgroup of patients with low back pain.

The aim of the study is to clarify whether proprioceptive training has a positive effect on proprioceptive postural control in individuals with recurrent low back pain.

ELIGIBILITY:
Inclusion Criteria individuals with low back pain:

* Age: 18-45 years old
* At least 1 year of low back pain with/without referred pain in buttock/thigh
* At least 3 episodes of disabling low back pain
* At least a score of 20% on the Oswestry Disability Index
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, multiple sclerosis, stroke, history of vestibular disorder, respiratory disease, pregnancy
* Radicular symptoms
* Not Dutch-speaking
* Strong opioids
* Neck pain
* Smoking history

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Proprioceptive postural control | 12 weeks
  Center of pressure displacement (force plate) in standing in response to local muscle vibration on ankle and back muscles to specifically detect the role of proprioception in postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, PhD, Principal Investigator — KU Leuven; Thierry Troosters, PhD, Principal Investigator — KU Leuven; Roeland Lysens, MD, PhD, Principal Investigator — KU Leuven; Peter Van Wambeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

REFERENCES:
- [Background] Claeys K, Brumagne S, Dankaerts W, Kiers H, Janssens L. Decreased variability in postural control strategies in young people with non-specific low back pain is associated with altered proprioceptive reweighting. Eur J Appl Physiol. 2011 Jan;111(1):115-23. doi: 10.1007/s00421-010-1637-x. Epub 2010 Sep 8. PMID 20824281
- [Background] Johanson E, Brumagne S, Janssens L, Pijnenburg M, Claeys K, Paasuke M. The effect of acute back muscle fatigue on postural control strategy in people with and without recurrent low back pain. Eur Spine J. 2011 Dec;20(12):2152-9. doi: 10.1007/s00586-011-1825-3. Epub 2011 May 1. PMID 21533851
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397
- [Background] Brumagne S, Janssens L, Knapen S, Claeys K, Suuden-Johanson E. Persons with recurrent low back pain exhibit a rigid postural control strategy. Eur Spine J. 2008 Sep;17(9):1177-84. doi: 10.1007/s00586-008-0709-7. Epub 2008 Jul 2. PMID 18594876
- [Background] Brumagne S, Janssens L, Janssens E, Goddyn L. Altered postural control in anticipation of postural instability in persons with recurrent low back pain. Gait Posture. 2008 Nov;28(4):657-62. doi: 10.1016/j.gaitpost.2008.04.015. Epub 2008 Jun 9. PMID 18541428
- [Derived] Janssens L, Brumagne S, Claeys K, Pijnenburg M, Goossens N, Rummens S, Depreitere B. Proprioceptive use and sit-to-stand-to-sit after lumbar microdiscectomy: The effect of surgical approach and early physiotherapy. Clin Biomech (Bristol). 2016 Feb;32:40-8. doi: 10.1016/j.clinbiomech.2015.12.011. Epub 2016 Jan 6. PMID 26795132